CLINICAL TRIAL: NCT06325982
Title: Clinical Observation of Trolamine Retention Enema in Preventing Acute Radiation-induced Rectal Injury: a Real-world Multicenter Prospective Study
Brief Title: Clinical Observation of Drug Retention Enema in Preventing Acute Radiation-induced Rectal Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BYFFL-01
Record Dates: First submitted 2024-03-11; First posted 2024-03-22 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Radiation Injuries; Rectal Diseases
MeSH Terms: conditions — Radiation Injuries; Rectal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triethanolamine cream group (Experimental): Triethanolamine cream retention enema was given once every night before going to bed during radiotherapy until the end of radiotherapy. Triethanolamine cream retention enema was given once before going to bed the day after radiotherapy for 3 months
  Interventions: Drug: Triethanolamine cream

INTERVENTIONS:
Drug: Triethanolamine cream — Triethanolamine cream retention enema was given once every night before going to bed during radiotherapy until the end of radiotherapy. Triethanolamine cream retention enema was given once before going to bed the day after radiotherapy for 3 months.
  Preparation method: Pull out the syringe piston, add 15ml triethanolamine cream, add 30ml normal saline, gently pat, shake well.
  Specific methods of retention enema: at night before going to bed, empty urine and feces, prepare enema liquid into the syringe, connect the special catheter, and insert the other end of the special catheter into the anus (the special catheter can be applied with lubricant such as tea oil before insertion). The patient remained prone and semi-seated. Use a special catheter, insert a special catheter about 15cm from the anus, and inject enteral liquid while withdrawing, so that the liquid is retained in the rectum; The above treatment was performed before bed and retained overnight.

SUMMARY:
The main objective of this study was to evaluate the efficacy and safety of drug retention enema for the prevention of acute radiation rectal injury in the real world.

DETAILED DESCRIPTION:
The study was a prospective, multicenter, real-world study with eligible patient data as of May 1, 2024. The prospective study was a continuous, multicenter study.

ELIGIBILITY:
Inclusion Criteria:

* There are clear indications for radiotherapy (pelvic radiotherapy or rectal radiotherapy) according to relevant guidelines;
* ECOG score 0-1;
* normal mind, clear consciousness;
* High compliance;
* Able to cooperate with the interviewer

Exclusion Criteria:

* Poor compliance, unwilling to participate or unable to cooperate with the interviewer;
* Patients with other intestinal diseases (such as Crohn's disease, rectal ulcer, anal fissure, anal fistula, hemorrhoids, etc.) and perianal diseases;
* serious heart, brain, liver, kidney disease;
* Long-term immune dysfunction;
* Pregnant or lactating women;
* Patients who terminate treatment for various reasons.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-11 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence time of acute and chronic radiation rectal injury | Up to approximately 4 months
  RTOG/EORTC criteria were used to evaluate the severity of acute and chronic radiation rectal injury. The time (days) of acute radiation rectal injury were evaluated and recorded
Evaluation of acute and chronic radiation rectal injury | Up to approximately 4 months
  RTOG/EORTC criteria were used to evaluate the severity of acute and chronic radiation rectal injury. The grading of acute radiation rectal injury were evaluated and recorded

SECONDARY OUTCOMES:
Clinical symptom assessment | Up to approximately 4 months
  Clinical symptoms were assessed using the Simple Clinical Colitis Activity Index (SCCAI) designed by the Inflammatory Bowel Disease Research Group at the Royal Free Hospital School of Medicine.
  SCCAI in this study included 6 items, with a total score of 0-16. The higher the score, the more severe the symptoms.
Quality of life assessment assessed by IBDQ | Up to approximately 4 months
  The quality of life index (IBDQ) was used to evaluate the quality of life of patients with inflammatory bowel disease.
  IBDQ included 32 questions in 4 aspects: intestinal symptoms (10), systemic symptoms (5), emotional ability (12) and social ability (5). Each question was divided into 7 grades, with a total score of 32-224 points. The higher the score, the better the quality of life. Scores above 177 indicate light, 176-121 indicate medium, and below 120 indicate heavy.

CONTACTS AND LOCATIONS:
Overall Officials: lingdong Shao, Bachelor, Study Chair — Fujian Cancer Hospital
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No